CLINICAL TRIAL: NCT06752590
Title: A Phase IIa, Randomized, Double-blind, Placebo Controlled, Parallel Group, Multi-center Trial to Evaluate the Efficacy and Safety of ONO-1110 in Patients With Fibromyalgia
Brief Title: A Clinical Study of ONO-1110 in Patients With Fibromyalgia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-1110-05; jRCT2031240522 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia
Keywords: ONO-1110; ONO-1110-05; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-1110 (Experimental): ONO-1110 tablets once a day
  Interventions: Drug: ONO-1110
- Placebo (Placebo Comparator): Placebo tablets once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-1110 — ONO-1110 tablets once a day
  Arms: ONO-1110
Drug: Placebo — Placebo tablets once daily
  Arms: Placebo

SUMMARY:
To Evaluate the Efficacy and Safety of ONO-1110 in Patients with Fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

* Japanese (both sexes)
* Outpatient
* Patients who are considered capable of understanding the study procedures and completing the pain diary and questionnaires appropriately by the investigator (sub-investigator)
* Patients who meet the American College of Rheumatology Fibromyalgia Criteria

Exclusion Criteria:

* Patients with inflammatory arthritis, infectious arthritis, or autoimmune disease
* Patients with pain other than FM that may affect assessments in this study
* Patients with a past history of or concurrent neurologic diseases that may affect assessments in this study
* Patients with a past history of or concurrent malignant tumor within 3 years
* Patients who are pregnant, nursing, or possibly pregnant, or intending to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in weekly mean of average pain score from baseline to Week 8 of the treatment period | Up to 16 weeks
Adverse events | Up to 16 weeks

SECONDARY OUTCOMES:
Change in weekly mean of average pain score from baseline in each week | Up to 16 weeks
30%- and 50%-responder rates based on the weekly mean of average pain score | Up to 16 weeks
  proportions of participants whose weekly mean of average pain score has decreased by 30% and 50% from baseline, respectively
Change in weekly mean of worst pain score from baseline to each week | Up to 16 weeks
30%- and 50%-responder rates based on the weekly mean of worst pain score | Up to 16 weeks
  proportions of participants whose weekly mean of worst pain score has decreased by 30% and 50% from baseline, respectively
Change in WPI and SSS score of 2016 Revised FM Diagnostic Criteria by ACR from baseline | Up to 16 weeks
Change in Japanese version of the Revised Fibromyalgia Impact Questionnaire (JFIQR) score from baseline | Up to 16 weeks
Change in Patient Global Impression of Change (PGIC) score from baseline | Up to 16 weeks
Change in Hospital Anxiety and Depression Scale (HADS) score from baseline | Up to 16 weeks
Change in Medical Outcomes Study Sleep Scale (MOS-Sleep Scale) score from baseline | Up to 16 weeks
Plasma ONO-1110 concentrations | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (27):
- Japan (27):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Kimura Clinic, Nagoya, Aichi-ken
  - National Hospital Organization Shimoshizu National Hospital, Yotsukaidō, Chiba
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Shirasawa Orthopedic Clinic, Morioka, Iwate
  - Kokorotoitami Clinic, Kawasaki, Kanagawa
  - Women's Clinic Luna, Yokohama, Kanagawa
  - Miyashita Rheumatology Clinic, Ōmura, Nagasaki
  - Medical Corporation Fujigaki Clinic, Ōita, Oita Prefecture
  - Ai Sakura Clinic, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Japanese Red Cross Okayama Hospital, Okayama
  - Hayaishi Hospital, Osaka
  - Morimoto Clinic, Osaka
  - Shizuoka Rehab Pain Clinic, Shizuoka
  - Fukuwa Clinic, Tokyo
  - Ginza Neurological Clinic, Tokyo
  - Himenotomomi Clinic, Tokyo
  - Ikebukuro Internal Medicine, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Tokyo
  - Juntendo University Hospital, Tokyo
  - Juntendo University Nerima Hospital, Tokyo
  - Nihonbashi Medical, Tokyo
  - Nishiogi Pain Clinic, Tokyo
  - Sanno Hospital, Tokyo
  - Tokyo-Eki Center-Building Clinic, Tokyo
  - Yakushinkai Healthcare Association Kandasudacho Dermatology, Tokyo

IPD SHARING:
Plan to Share IPD: No